CLINICAL TRIAL: NCT01405651
Title: A Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-6950 in Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-6950 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-6950POU002
Record Dates: First submitted 2011-07-22; First posted 2011-07-29 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Adult Subjects
Keywords: ONO-6950; Healthy adult subjects
MeSH Terms: interventions — gemilukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- E (Experimental): ONO-6950
  Interventions: Drug: ONO-6950
- P (Placebo Comparator): Placebo
  Interventions: Drug: ONO-6950

INTERVENTIONS:
Drug: ONO-6950 — 30 mg, 100 mg, 300 mg at multiple doses
  Arms: E
Drug: ONO-6950 — Placebo to match ONO-6950 tablets dosed in a similar manner to ONO-6950
  Arms: P

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of ONO-6950 across ascending multiple doses in healthy adult male and female subjects. The secondary objectives are to characterize the PK and pharmacodynamic (PD) profiles of ONO-6950 by measuring plasma concentrations of ONO-6950 and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male or female subjects (18-55 inclusive)
* Body mass index (BMI)of 10-35 kg/m2 (inclusive)
* For females; postmenopausal, non-lactating, and non-pregnant

Exclusion Criteria:

* History or presence of clinical significant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-6950 using vital signs, pulmonary function tests ECGs, laboratory tests and physical examinations | At protocol-specified timepoints before and after study drug administration up to 21 days

SECONDARY OUTCOMES:
Characterization of PK ( Cmax, Tmax, AUC, ty2, etc.) and PD profiles of ONO-6950 using plasma concentration of ONO-6950 in blood and pulmonary function tests | At protocol-specified timepoints before and after study drug administration up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (1):
- Miramar Clinical Site, Miramar, Florida, United States